CLINICAL TRIAL: NCT03534856
Title: Pilot Study of Sensorimotor Changes in Stroke Following Mindfulness
Brief Title: Sensorimotor Changes in Stroke Following Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sook-Lei Liew, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS1500196C0005
Record Dates: First submitted 2018-04-17; First posted 2018-05-23 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Spasticity, Muscle
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness meditation (Experimental): Two weeks of short, daily guided mindfulness meditations were provided.
  Interventions: Behavioral: Mindfulness meditation

INTERVENTIONS:
Behavioral: Mindfulness meditation — Short guided mindfulness meditations were provided on an MP3 player.

SUMMARY:
Roughly 30% of stroke survivors experience spasticity, a velocity-dependent increase in stretch reflexes. In this pilot study, the investigators aimed to examine the effects of mindfulness meditation on spasticity and quality of life in individuals after stroke.

DETAILED DESCRIPTION:
Thirty percent of stroke survivors experience spasticity, a velocity dependent increase in stretch reflexes, which negatively affects quality of life and activities of daily living (Thibaut et al. 2013). Spasticity is a secondary neurological symptom induced by neurological hyperreflexia seen in stroke and other neurological disorders (Bose et al. 2015). If left untreated, stroke survivors may develop contractures which can further impede motor recovery and participation in activities of daily life (Thibaut et al. 2013). Spasticity is typically treated with medications, botox injections, baclofen intrathecal pumps, occupational therapy, and physical therapy, but current treatment options are often expensive and effectiveness is generally unsatisfactory (Kheder and Nair 2012). Thus, there is a need to find low-cost, effective, and accessible methods that have the potential to help reduce spasticity and promote recovery.

Increased spasticity has been linked to emotion-based stress, such as anxiety (Bhimani and Anderson 2014). Previous research has anecdotally linked meditation, a technique that has been used to reduce anxiety, to decreased post-stroke spasticity (Bhimani and Anderson 2014). In this pilot study, the researchers aimed to test whether two weeks of mindfulness meditation could lead to reduced anxiety and reduced post-stroke spasticity. Briefly, mindfulness meditation is a type of meditation that trains awareness and acceptance of the current inner and outer reality, and is often taught through Jon Kabat-Zinn's 8-week Mindfulness Based Stress Reduction (MBSR) course (Kabat-Zinn 1996). Importantly, while it is typically taught by an experienced teacher over a series of sessions, studies have also shown successful mindfulness practice via audio/video recording (Potter 2017), allowing for greater accessibility to mindfulness training for broader audiences, including those with mobility limitations.

Although studies have found that mindfulness meditation may be linked to mood, anxiety, and pain reduction, it has not been directly connected to motor function or spasticity (Creswell et al. 2014; Moustgaard et al. 2007; Zeidan et al. 2010). Specifically, mindfulness intervention studies have reported decreased mental fatigue in people with TBI or stroke (Johansson et al. 2012) and a reduction in psychological stress and improvement in cognitive function in patients with multiple sclerosis (Blankespoor et al. 2017). One systematic review showed that mindfulness meditation helped patients cope with their chronic illnesses, including cancer, depression and general anxiety disorder, by improving their mood and anxiety symptoms (Hofmann et al. 2010). In stroke and transient ischemic attack survivors, there is small but growing evidence that mindfulness promotes positive results for psychological and psychosocial health (Lawrence et al. 2013). A pilot study with individuals after stroke used an 8-week Mindfulness-Based Cognitive Therapy (MBCT) intervention, which is a combination of MBSR with some insights from cognitive behavioral therapy, and found a reduction in anxiety and depression and an increase in quality of life, including physical functioning. (Moustgaard et al. 2007).

Because of the anecdotal evidence linking stress to increased spasticity and the clinical evidence linking meditation to decreased stress, the researchers conducted a pilot study to explore whether two weeks of guided mindfulness meditation-a low-cost, home-based intervention-could improve spasticity, along with quality of life, stress and anxiety, in individuals after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke (greater than 1 year post stroke)
* Over 18 years old
* Moderate to severe motor deficits with self-reported spasticity
* No prior mindfulness meditation experience

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Modified Ashworth Scale at 2 weeks | This was measured before and after two weeks of meditation
  This scale measures post-stroke spasticity on a scale that ranges from 0-4 where 0 is no spasticity and the higher value represents a greater spasticity

SECONDARY OUTCOMES:
Change from Baseline Fugl Meyer Upper Extremity Scale at 2 weeks | This was measured before and after two weeks of meditation
  This is a measure of sensory and motor impairment after stroke. This scale ranges from 0 - 66, where 0 represents greater impairment and 66 represents no impairment.
Change from Baseline Stroke Specific Quality of Life Survey at 2 weeks | This was measured before and after two weeks of meditation
  This is a quality of life survey for individuals after stroke, with the following subscales:
  i. Mobility (Range: 0-30), higher values represent a better outcome ii. Energy (Range: 0-15), higher values represent a better outcome iii. Upper Extremity Function (Range: 0-25), higher values represent a better outcome iv. Work/productivity (Range: 0-15), higher values represent a better outcome v. Mood (Range: 0-25), higher values represent a better outcome vi. Self-care (Range: 0-25), higher values represent a better outcome vii. Social Roles (Range: 0-25), higher values represent a better outcome viii. Family Roles (Range: 0-15), higher values represent a better outcome ix. Vision (Range: 0-15), higher values represent a better outcome x. Language (Range: 0-25), higher values represent a better outcome xi. Thinking (Range: 0-15), higher values represent a better outcome xii. Personality (Range: 0-15), higher values represent a better outcome
Change from Baseline Freiburg Mindfulness Inventory at 2 weeks | This was measured before and after two weeks of meditation
  This measure is of self-reported mindfulness capacity. Scores range from 14-56, where higher scores represent greater mindfulness ability.
Change from Baseline Hospital Anxiety and Depression Scale at 2 weeks | This was measured before and after two weeks of meditation
  This is an assessment of anxiety and depression. There are two subscales - i. Anxiety Subscale (Range: 0-21), higher values represent a worse outcome ii. Depression Subscale (Range: 0-21), higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wathugala M, Saldana D, Juliano JM, Chan J, Liew SL. Mindfulness Meditation Effects on Poststroke Spasticity: A Feasibility Study. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X19855941. doi: 10.1177/2515690X19855941. PMID 31215234